CLINICAL TRIAL: NCT04404439
Title: Treatment of Tinnitus With Migraine Medications: A Randomized Clinical Trial
Brief Title: Treatment of Tinnitus With Migraine Medications
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of California, Irvine (Other)
Responsible Party: Principal Investigator, Hamid Djalilian, Professor, Neurotology and Skull Base Surgery, University of California, Irvine
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HS# 2018-4458
Record Dates: First submitted 2020-05-17; First posted 2020-05-27 (Actual); Last update posted 2023-01-09 (Actual); Status verified 2023-01

CONDITIONS: Tinnitus, Subjective; Tinnitus
Keywords: tinnitus; medication; randomized; RCT; trial; migraine
MeSH Terms: conditions — Tinnitus; Migraine Disorders | interventions — Nortriptyline; Topiramate; Verapamil; Paroxetine

STUDY DESIGN:
Intervention Model Description: Participants will be assigned to a study group by chance (like a coin flip) rather than by a medical decision made by the researchers. There are three arms in the study (treatment group 1 which consists of nortriptyline + topiramate, treatment group 2 which consist of verapamil + paroxetine, and a placebo group), and participants enrolling in the trial will be randomly assigned in a 1:1:1 fashion to one of the arms. The participant will remain in the same arm for the duration of the study (8 weeks). There may be multiple participants in each arm who are undergoing the study at the same time (parallel model).
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Nortriptyline + topiramate (Experimental): Nortriptyline (7.5 mg) plus topiramate (10 mg) in a single pill initially taken once daily. Dose may be increased as directed by care provider by 7.5mg weekly (to a maximum of 60mg) for nortriptyline, and by 10mg weekly (maximum 80mg) for topiramate.
  Interventions: Drug: Nortriptyline + topiramate
- Verapamil + paroxetine (Experimental): Verapamil (30 mg) plus paroxetine (4 mg) in a single pill initially taken once daily. Dose may be increased as directed by care provider by 30mg weekly (to a maximum of 240mg) for verapamil, and by 4mg weekly (maximum 32mg) for paroxetine.
  Interventions: Drug: Verapamil + paroxetine
- Placebo (Placebo Comparator): Placebo pill.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Nortriptyline + topiramate — Treatment group 1
  Arms: Nortriptyline + topiramate
Drug: Verapamil + paroxetine — Treatment group 2
  Arms: Verapamil + paroxetine
Other: Placebo — Placebo comparator
  Arms: Placebo

SUMMARY:
Tinnitus represents one of the most common and distressing otologic problems, and it causes various somatic and psychological disorders that interfere with the quality of life. It is well-understood that many factors, such as poor education, lower income, or occupational, and recreational activity associated with high noise exposure, influences the prevalence and risk of tinnitus. Although the economic and emotional impact of tinnitus is large, there is currently no FDA-approved medication to treat this condition. However, there are pharmacological options to address the stress, anxiety, and depression that are caused by tinnitus. In this project, we intend to use medications for patients with tinnitus in order to decrease the impact of tinnitus on their daily life and activities.

DETAILED DESCRIPTION:
This study is 8 weeks in duration. There are three arms in the experiment: the first is nortriptyline (7.5 mg) plus topiramate (10 mg), the second is verapamil (30 mg) plus paroxetine (4 mg), and the third is a placebo group. This is a double-blinded trial. Participants will be randomized to one arm for the duration of the trial using simple randomization with a computer-generated number. Both medication combinations and placebo may include dosage increases weekly if symptoms do not improve. Nortriptyline may be increased by 7.5mg weekly (to a maximum of 60mg), topiramate by 10mg weekly (maximum 80mg), verapamil by 30mg weekly (maximum 240mg), and paroxetine by 4mg weekly (maximum 32mg). Symptomatic survey scores from each arm will be obtained before and after treatment and weekly. An unblinded neurotologist attending (Dr. Harrison Lin) will also become involved with patients' treatments as they start to report changes in symptoms in order to monitor their safety and provide advice on change in dosage if patients have questions.

ELIGIBILITY:
Inclusion Criteria:

* Patients with moderate to severe tinnitus.
* Male or female between the ages of 25 to 85 years.
* Subject must be compliant with the medication and attend study visits.
* Must be able to read and write in the English language to provide consenting.

Exclusion Criteria:

* Pregnancy will result in automatic exclusion from the study. Rule out of pregnancy will be done by a urine pregnancy test to confirm the situation for all women who are of child bearing potential.
* Subject with history of an adverse reaction to medication being prescribed.
* Subject suffers from a medical condition or has history that may be concerning to the investigators clinical opinion.
* All contraindications for the medications which prevent subjects from randomization will be considered as exclusion criteria.

Ages: 25 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2019-09-26 (Actual); Primary Completion 2023-12-30 (Estimated); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
Tinnitus Functional Index (TFI) | 8 weeks
  Subjective improvement from baseline in tinnitus symptoms as measured by Tinnitus Functional Index (TFI). The TFI is scored from 0% to 100%, with higher scores indicating a more negative impact of tinnitus.

SECONDARY OUTCOMES:
Visual Analog Scale (VAS) | 8 weeks
  Subjective improvement in tinnitus loudness severity based on a visual analog scale (VAS). The VAS is scored from 0 to 10, with a higher score representing an increased severity of tinnitus.
Patient Health Questionnaire (PHQ) | 8 weeks
  Subjective improvement in depression symptoms based on patient health questionnaire (PHQ). The PHQ is scored from 0 to 27, with a higher score indicating increased depression severity.
Perceived Stress Scale (PSS) | 8 weeks
  Subjective improvement in stress based on perceived stress scale (PSS). The PSS is scored from 0 to 40, with higher scores indicating higher perceived stress.
Sleep Quality Index (SQI) | 8 weeks
  Subjective improvement in sleep quality based on sleep quality index (SQI). The SQI is scored from 0 to 21, with higher scores indicating worse quality of sleep.

CONTACTS AND LOCATIONS:
Overall Officials: Hamid R Djalilian, MD, Principal Investigator — Univeristy of California, Irvine
Locations (1):
- University of California, Irvine Medical Center ENT Clinic (Pavilion 2), Orange, California, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Evans RW, Ishiyama G. Migraine with transient unilateral hearing loss and tinnitus. Headache. 2009 May;49(5):756-8. doi: 10.1111/j.1526-4610.2008.01075.x. No abstract available. PMID 19472451
- [Background] Sindhusake D, Golding M, Newall P, Rubin G, Jakobsen K, Mitchell P. Risk factors for tinnitus in a population of older adults: the blue mountains hearing study. Ear Hear. 2003 Dec;24(6):501-7. doi: 10.1097/01.AUD.0000100204.08771.3D. PMID 14663349
- [Background] Dobie RA. A review of randomized clinical trials in tinnitus. Laryngoscope. 1999 Aug;109(8):1202-11. doi: 10.1097/00005537-199908000-00004. PMID 10443820
- [Background] Langguth B, Hund V, Busch V, Jurgens TP, Lainez JM, Landgrebe M, Schecklmann M. Tinnitus and Headache. Biomed Res Int. 2015;2015:797416. doi: 10.1155/2015/797416. Epub 2015 Oct 25. PMID 26583133
- [Background] Langguth B, Hund V, Landgrebe M, Schecklmann M. Tinnitus Patients with Comorbid Headaches: The Influence of Headache Type and Laterality on Tinnitus Characteristics. Front Neurol. 2017 Aug 28;8:440. doi: 10.3389/fneur.2017.00440. eCollection 2017. PMID 28894434
- [Background] Guichard E, Montagni I, Tzourio C, Kurth T. Association Between Headaches and Tinnitus in Young Adults: Cross-Sectional Study. Headache. 2016 Jun;56(6):987-94. doi: 10.1111/head.12845. Epub 2016 May 20. PMID 27197786
- [Background] Duckert LG, Rees TS. Treatment of tinnitus with intravenous lidocaine: a double-blind randomized trial. Otolaryngol Head Neck Surg. 1983 Oct;91(5):550-5. doi: 10.1177/019459988309100514. PMID 6417606
- [Background] Hallam RS, McKenna L, Shurlock L. Tinnitus impairs cognitive efficiency. Int J Audiol. 2004 Apr;43(4):218-26. doi: 10.1080/14992020400050030. PMID 15250126
- [Background] Muhlau M, Rauschecker JP, Oestreicher E, Gaser C, Rottinger M, Wohlschlager AM, Simon F, Etgen T, Conrad B, Sander D. Structural brain changes in tinnitus. Cereb Cortex. 2006 Sep;16(9):1283-8. doi: 10.1093/cercor/bhj070. Epub 2005 Nov 9. PMID 16280464
- [Background] Landgrebe M, Langguth B, Rosengarth K, Braun S, Koch A, Kleinjung T, May A, de Ridder D, Hajak G. Structural brain changes in tinnitus: grey matter decrease in auditory and non-auditory brain areas. Neuroimage. 2009 May 15;46(1):213-8. doi: 10.1016/j.neuroimage.2009.01.069. Epub 2009 Feb 12. PMID 19413945
- [Background] Price JL, Drevets WC. Neurocircuitry of mood disorders. Neuropsychopharmacology. 2010 Jan;35(1):192-216. doi: 10.1038/npp.2009.104. PMID 19693001
- [Background] Ploghaus A, Tracey I, Gati JS, Clare S, Menon RS, Matthews PM, Rawlins JN. Dissociating pain from its anticipation in the human brain. Science. 1999 Jun 18;284(5422):1979-81. doi: 10.1126/science.284.5422.1979. PMID 10373114
- [Background] Wager TD, Rilling JK, Smith EE, Sokolik A, Casey KL, Davidson RJ, Kosslyn SM, Rose RM, Cohen JD. Placebo-induced changes in FMRI in the anticipation and experience of pain. Science. 2004 Feb 20;303(5661):1162-7. doi: 10.1126/science.1093065. PMID 14976306
- [Background] Roberts LE, Eggermont JJ, Caspary DM, Shore SE, Melcher JR, Kaltenbach JA. Ringing ears: the neuroscience of tinnitus. J Neurosci. 2010 Nov 10;30(45):14972-9. doi: 10.1523/JNEUROSCI.4028-10.2010. PMID 21068300
- [Background] Minen MT, Camprodon J, Nehme R, Chemali Z. The neuropsychiatry of tinnitus: a circuit-based approach to the causes and treatments available. J Neurol Neurosurg Psychiatry. 2014 Oct;85(10):1138-44. doi: 10.1136/jnnp-2013-307339. Epub 2014 Apr 17. PMID 24744443
- [Background] Llinas RR, Ribary U, Jeanmonod D, Kronberg E, Mitra PP. Thalamocortical dysrhythmia: A neurological and neuropsychiatric syndrome characterized by magnetoencephalography. Proc Natl Acad Sci U S A. 1999 Dec 21;96(26):15222-7. doi: 10.1073/pnas.96.26.15222. PMID 10611366
- [Background] Muhlnickel W, Elbert T, Taub E, Flor H. Reorganization of auditory cortex in tinnitus. Proc Natl Acad Sci U S A. 1998 Aug 18;95(17):10340-3. doi: 10.1073/pnas.95.17.10340. PMID 9707649